CLINICAL TRIAL: NCT07393854
Title: Clinical Success and Parental Satisfaction of Two Commercially Available Stainless Steel Crowns in Pediatric Patients Under General Anesthesia: A Comparative Study
Brief Title: Clinical Success of Two Stainless Steel Crowns in Children Treated Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Narmin Mammadli, Principal Investigator, Bezmialem Vakif University
Other Study IDs: 08.06.2023-E.110543
Record Dates: First submitted 2026-01-27; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Dental Caries; General Anesthesia; Pediatric Dentistry
Keywords: steenless steel crown; pediatric dental treatments; general anesthesia; restorative dental treatments
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Nu Smile Group: This group consists of pediatric patients aged 2-8 years who have received Nu Smile stainless steel crowns under general anesthesia at Bezmialem Vakıf University Faculty of Dentistry. Participants have a minimum postoperative period of 6 months and will be evaluated based on clinical success and parental satisfaction.
  Interventions: Device: NuSmile Stainless Steel Crown
- Kids Crown Group: This group consists of pediatric patients aged 2-8 years who have received Kids Crown stainless steel crowns under general anesthesia at Bezmialem Vakıf University Faculty of Dentistry. Participants have a minimum postoperative period of 6 months and will be evaluated based on clinical success and parental satisfaction.
  Interventions: Device: Kids Crown Stainless Steel Crown

INTERVENTIONS:
Device: NuSmile Stainless Steel Crown — NuSmile stainless steel crowns were placed as part of routine pediatric dental treatment under general anesthesia. The crowns were placed at least 6 months prior to study evaluation. No intervention is applied during the study period; outcomes are assessed retrospectively at follow-up.
  Groups: Nu Smile Group
Device: Kids Crown Stainless Steel Crown — Kids Crown stainless steel crowns were placed as part of routine pediatric dental treatment under general anesthesia. The crowns were placed at least 6 months prior to study evaluation. No intervention is applied during the study period; outcomes are assessed retrospectively at follow-up.
  Groups: Kids Crown Group

SUMMARY:
The purpose of this study is to compare the clinical performance and parental satisfaction of two commercially available stainless steel crown systems used in pediatric patients treated under general anesthesia. Children aged 2-8 years who received at least one stainless steel crown under general anesthesia with a minimum follow-up period of 6 months will be evaluated.

Clinical outcomes will include crown retention, occlusal contact, gingival health, and other crown-related parameters assessed during follow-up examinations. Parental satisfaction regarding aesthetics, function, durability, and overall acceptance of the crowns will be assessed using a structured questionnaire.

DETAILED DESCRIPTION:
This observational clinical study is designed to compare the clinical performance and parental satisfaction of two commercially available stainless steel crown systems (NuSmile and Kids Crown) placed in pediatric patients treated under general anesthesia.

The study population consists of children aged 2-8 years who received at least one stainless steel crown under general anesthesia at the Department of Pediatric Dentistry, Bezmialem Vakıf University, within the previous three years. Only restorations with a minimum postoperative follow-up of 6 months will be evaluated. All clinical examinations will be completed during a defined 1-month assessment period.

Clinical evaluations will be performed by a single calibrated examiner to ensure consistency and reduce inter-examiner variability. Examinations will be conducted under standardized dental light conditions using a dental mirror and curved explorer. A structured and previously validated scoring system adapted from the literature will be applied for all clinical assessments.

The clinical evaluation will focus on crown-related outcomes, including retention, occlusal contact, proximal contact adaptation, crown integrity, gingival response, and oral hygiene status. Additional clinical signs such as pain, swelling, fistula formation, percussion sensitivity, and tooth mobility will also be recorded to identify potential biological or functional complications associated with the restorations.

Parental satisfaction will be assessed using a structured questionnaire administered to parents or legal guardians at the follow-up visit. Satisfaction will be evaluated using a 5-point Likert scale addressing aesthetic appearance, functional performance, durability, and overall acceptance of the stainless steel crowns.

Statistical analyses will be conducted to compare clinical outcomes and parental satisfaction between the two crown systems. Appropriate statistical tests will be selected based on data distribution and variable characteristics, with statistical significance set according to conventional thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-8 years
* Have received at least one stainless steel crown restoration under general anesthesia at Bezmialem Vakıf University Faculty of Dentistry
* Have a minimum postoperative period of 6 months
* Parents provided written informed consent

Exclusion Criteria:

* Children whose parents did not provide written consent
* Children with chronic systemic diseases
* Children with physical or mental disabilities

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will include pediatric patients aged 2-8 years who have previously undergone stainless steel crown restorations under general anesthesia. Only patients with a minimum postoperative period of 6 months will be included. The study aims to evaluate clinical success and parental satisfaction regarding these restorations.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Overall Clinical Success of Stainless Steel Crowns (Composite Outcome) | 1 month (single follow-up assessment for all participants with a minimum of 6 months postoperative period)
  Overall clinical success will be defined as the presence of a clinically acceptable stainless steel crown at follow-up, based on a composite assessment of predefined clinical parameters. A crown will be considered clinically successful only if all criteria listed below are met.
  Clinical success criteria include:
  Crown retention (present) Occlusal contact (present) Proximal contact adaptation (acceptable) Absence of crown perforation Absence of pain or swelling Absence of fistula formation Absence of tenderness to percussion Absence of pathological tooth mobility Gingival health score ≤1 on the Gingival Index
  Unit of Measure:
  Binary outcome (Successful / Unsuccessful)

SECONDARY OUTCOMES:
Gingival Health Around Stainless Steel Crowns | 1 month (single clinical assessment at follow-up visit)
  Gingival health will be assessed using the Gingival Index (Löe and Silness) to evaluate inflammation of the gingival tissues adjacent to the crowns.
  Scale:
  Gingival Index (GI):
  0 = Normal gingiva
  1. = Mild inflammation
  2. = Moderate inflammation
  3. = Severe inflammation Higher scores indicate worse gingival health.
Parental Satisfaction with Stainless Steel Crowns | 1 month (single questionnaire-based assessment at follow-up visit)
  Parental satisfaction will be assessed using a structured questionnaire based on a 5-point Likert scale, evaluating parental perception of the stainless steel crowns.
  Domains assessed include:
  Aesthetic satisfaction (color, appearance, shape, size) Functional satisfaction (durability, retention, comfort) Overall acceptance and parental preference
  Scale:
  5-point Likert scale (1 = very dissatisfied, 5 = very satisfied) Higher scores indicate greater parental satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Başak Günay, DDS, Study Director — Bezmialem Vakıf University Faculty of Dentistry
Locations (1):
- Bezmialem Vakıf University Faculty of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and ethical considerations related to patient confidentiality.